CLINICAL TRIAL: NCT05152251
Title: Investigation of Activity and Participation Levels in Children With Down Syndrome
Brief Title: Activities and Participation of Children With Down Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Duygu Turker, Assistant Professor, Hacettepe University
Other Study IDs: 2021-365
Record Dates: First submitted 2021-11-29; First posted 2021-12-09 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Down Syndrome; Activity; Participation; Quality of Life
MeSH Terms: conditions — Down Syndrome; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Down Syndrome
  Interventions: Other: Evaluation
- Control Group: Typically Developing Children
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — Individuals' activity participation levels and the restrictive or supportive factors affecting their participation levels and their effects on quality of life will be evaluated.

SUMMARY:
The aim of this study is to examine the activity participation levels of Down syndrome(DS) children and the restrictive or supportive factors affecting their participation levels and to investigate their effects on quality of life. 35 children diagnosed with DS by a pediatric neurologist and 35 typically developing children are planned to be included in this study. Sociodemographic data of typically developing and DS children who agreed to participate in the study and their families will be questioned. Activity (Gross Motor Function Measurement-GMFM-88) , participation and the effect of the environment on participation (Participation and Environment Measure for Children and Youth-PEM-CY ), reflection of motor development levels to functions in daily living activities (Pediatric Evaluation of Disability Inventory- PEDI) , quality of life(Pediatric Quality of Life Inventory- PedsQL) and familial impact (Impact on Family Scale-IPFAM) will be evaluated. Evaluation methods to be used in our study will be applied one-on-one with children and face-to-face interviews with their parents. Our study is important in that there is little evidence on participation studies in children and that changing medical paradigms emphasize the quality of life of children. In addition, the PEM-CY the investigators will use in the study will make the study more valuable as it examines the effect of the environment on participation and evaluates participation in different environments.

DETAILED DESCRIPTION:
The aim of this study is to examine the activity participation levels of DS children and the restrictive or supportive factors affecting their participation levels and to investigate their effects on quality of life. 35 children diagnosed with DS by a pediatric neurologist and 35 typically developing children are planned to be included in this study. In line with the power analysis, a study should be conducted with a total of 52 individuals, 26 individuals in each group, with 95% confidence (1-α), 95.0% test power (1-β) and d=1.50 (large) effect size . Considering the 25% loss of individuals in the groups during the evaluation period, it was decided that forming each group with at least 35 children would increase the power of the study, and the study will be concluded with at least 70 individuals.Sociodemographic data of typically developing and DS children who agreed to participate in the study and their families will be questioned. Sociodemographic data will include information about age, height, weight, gender, body mass index, education level of the child, place of residence, physical therapy and special education session received by the child, assistive devices used, comorbidities of the child (cardiovascular anomalies, pulmonary problems, oral disorders, gastrointestinal disorders, overweight and obesity, musculoskeletal disorders, epilepsy), age of parents, education level, occupation, marital status, average income . Activity (Gross Motor Function Measurement-GMFM-88) , participation and the effect of the environment on participation (Participation and Environment Measure for Children and Youth -PEM-CY), reflection of motor development levels to functions in daily living activities (Pediatric Evaluation of Disability Inventory- PEDI) , quality of life(Pediatric Quality of Life Inventory- PedsQL) and familial impact (Impact on Family Scale-IPFAM) will be evaluated. Evaluation methods to be used in our study will be applied one-on-one with children and face-to-face interviews with their parents. The data to be obtained from the study will be analyzed using appropriate statistical methods. Statistical analyzes will be made using the Windows compatible Statistical Package for Social Science(SPSS) 20.0 package program. Data indicated by measurement will be expressed as arithmetic mean and standard deviation, data indicated by counting will be expressed as n and percentage (n,%). In the comparison of the groups, the t test will be used when parametric conditions are met, and the Mann Whitney U test will be used in cases where they are not met. The P value will be taken as 0.05. The investigators think that the results of the study can provide a new perspective to clinicians and researchers working in the field of rehabilitation in order to support the participation of DS children and young people in social life and can support social support projects and policies.

ELIGIBILITY:
Inclusion Criteria:

* Children with DS aged 8-17 years, who can cooperate, who have no visual and/or hearing impairment
* Typical developing children aged 8-17 years who are not diagnosed with any disease
* Parents who can read and write

Exclusion Criteria:

* Children and their families who did not want to participate in the study

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will include children with DS between the ages of 8-17, who can cooperate, who are not visually and/or hearing impaired, and typically developing children between the ages of 8-17 who are not diagnosed with any disease, and their literate parents.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measurement-88(GMFM-88) | The measurements will start with the first child with DS (estimated in November 2021) and will end with the evaluation of the 35th child(estimated in May 2022).
  The measurement assesses gross motor functions in children aged 5 months to 16 years.Although GMFM-88 was developed for children with Cerebral palsy (CP), it has also been validated for other populations such as children with DS and acquired brain injury.GMFM-88 consists of 88 items in total, including supine-prone position and rolling (A=17), sitting (B=20), crawling-kneeling (C=14), standing (D=13), walking-running-jumping (E=24) subsections. Gross motor functions in these items are evaluated according to the degree of achievement. Scoring is done according to the Likert scale: 0 means that the activity has never been started, and 3 means that 90% - 100% of the activity can be done.
Participation and Environment Measure for Children and Youth(PEM-CY) | The measurements will start with the first child (estimated in November 2021) and will end with the evaluation of the 70th child(estimated in May 2022).
  The PEM-CY is a parent report questionnaire used to assess participation and environmental factors in children and adolescents aged 5-17 years at home, at school, and in community settings. Items for each environment generally represent the types of activities performed in that setting; The engagement sections include 10 activities in the home environment, 5 activities in the school environment, and 10 activities in the community setting.For each type of activity, the parent is asked to rate how often (for the last 4 months) the child participates (eight options: daily to never), how much the child is typically involved during participation on a 5-point Likert scale, and whether the parent would like to see the child participate in this type of activity change.After answering the participation section, parents are asked to rate environmental features to identify supports and barriers.
Pediatric Evaluation of Disability Inventory(PEDI) | The measurements will start with the first child with DS (estimated in November 2021) and will end with the evaluation of the 35th child(estimated in May 2022).
  PEDI comprehensively assesses functional ability and performance in children with disabilities. The functional skills section, which measures the functional abilities of the child, consists of a total of 197 items including the Self-Care (73), Mobility (59) and Social Function (65) subscales. Rating 0; cannot and 1; is done as can be done. At the end of each sub-scale, the scores of that scale are summed up and the Functional Skills Total Score is obtained by adding the scores of the sub-scales.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory(PedsQL) | The measurements will start with the first child (estimated in November 2021) and will end with the evaluation of the 70th child(estimated in May 2022).
  It is a general quality of life scale that evaluates the physical and psychosocial lives of children between the ages of 2-18 independently of the disease. The scale, prepared for the 8-12 and 13-18 age groups, has a parent and child form. Scoring of the 23-item scale, which is suitable for use in both healthy and diseased children and adolescents, is done in 3 areas (total score, physical health, emotional social school functionality). The higher the total score, the better the health-related quality of life is perceived.
Impact on Family Scale(IPFAM) | The measurements will start with the first child with DS (estimated in November 2021) and will end with the evaluation of the 35th child(estimated in May 2022).
  It was developed to easily measure the impact on the families of children with chronic disabilities. It evaluates the level of influence of the family under 4 main headings: financial burden, familial and social impact, personal difficulty, coping, and the total impact score can be calculated by the sum of these parameters. The scale has a 4-point Likert type evaluation. A minimum of 24 and a maximum of 96 points can be obtained from the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Türker, PhD,PT, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Health Sciences University, Ankara, Turkey (Türkiye)